CLINICAL TRIAL: NCT05343442
Title: A Novel Technique for Safe Blind Percutaneous Tracheostomy
Brief Title: Percutaneous Tracheostomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0305355
Record Dates: First submitted 2022-04-13; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2021-11

CONDITIONS: Tracheostomy
Keywords: Intensive care unit; Trachea; Tracheostomy; Tracheostomy cannula; Critically ill
MeSH Terms: conditions — Tracheal Diseases; Critical Illness

STUDY DESIGN:
Intervention Model Description: Observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients assigned to percutaneous tracheostomy (Experimental): Guidewire dilating forceps (Grigges') technique was the method which has been applied during our work. Proper positioning: patient's neck was extended as much as possible by placing a rolled towel between the shoulder blades, the patient's neck and the bed were maintained in neutral position. The operative site was sterilized before draping with 10% povidone iodine solution. Lidocaine 2% was used as local anesthetic prior to beginning the intervention.
  Transverse (1 cm) skin incision was made midway between the cricoid cartilage and the suprasternal notch, i.e., opposite the 2nd - 3rd or 3rd - 4th tracheal rings. Blunt dissection of subcutaneous fat and pre-tracheal tissue with mosquito clamp in a vertical direction was done till the tracheal rings were palpable.
  Interventions: Procedure: Percutaneous tracheostomy

INTERVENTIONS:
Procedure: Percutaneous tracheostomy — Guidewire dilating forceps (Grigges') technique was the method which has been applied during our work. Proper positioning: patient's neck was extended as much as possible by placing a rolled towel between the shoulder blades, the patient's neck and the bed were maintained in neutral position. The operative site was sterilized before draping with 10% povidone iodine solution. Lidocaine 2% was used as local anesthetic prior to beginning the intervention.
  Transverse (1 cm) skin incision was made midway between the cricoid cartilage and the suprasternal notch, i.e., opposite the 2nd - 3rd or 3rd - 4th tracheal rings. Blunt dissection of subcutaneous fat and pre-tracheal tissue with mosquito clamp in a vertical direction was done till the tracheal rings were palpable.

SUMMARY:
Description of a technical modification of percutaneous tracheostomy that involves a safety method for confirming the intratracheal location of the needle at the time of puncture, with preventing serious complications such as false passage or damage to the posterior tracheal wall, without coadjuvant technique

DETAILED DESCRIPTION:
Introduction:

Tracheotomy is one of the most common procedures used in the Intensive Care Unit (ICU). Since 1985, percutaneous tracheotomy (PT) has gained widespread acceptance as a method for creating a surgical airway, and new techniques for PT have been developed. Furthermore, the technique could be performed at the patient bedside, leading to a new way of viewing surgical access to the airway in the critically ill patient.

In 1985, Ciaglia described percutaneous dilatational tracheotomy (PDT). Five years later Griggs introduced tracheotomy using guidewire dilating forceps (GWDF). With this technique, the tracheostoma is opened using blunt-tipped forceps previously advanced over the metal guide in the tracheal lumen. In 1998 the classical technique of Ciaglia was modified using a single dilator with respect to the original technique, this modification offered the advantage that the stoma is produced by a single dilatation, thereby avoiding the need for successive dilatations.

PDT heralds many peri-procedural complications as bleeding, difficulty to place the tube, false passage, posterior tracheal wall injury, pneumothorax, pneumomediastinum, and subcutaneous emphysema. In view of preventing serious complications, fibro-bronchoscopy is the most widely used safety method, though its application as a routine coadjuvant technique is a subject of controversy, since the endoscopic guide produces a rise in airway pressure, hypoventilation, and an increase in intracranial pressure; a situation that contraindicates its utilization in some patients. Moreover, bronchoscopy increases the cost of the procedure. Capnography is useful for confirming the intratracheal location of the needle at the time of puncture. The disadvantage of capnography is the lack of direct visualization of the precise position of the needle and metal guide within the trachea. Ultrasound is a noninvasive procedure and can be useful for locating aberrant vascular structures.

One of the main advantages of percutaneous tracheotomy is bedside performance, thus eliminating the hazards, expenses, and logistics involved in operating room set-up usually required for open surgical tracheotomies. So, searching for a safe way without coadjuvant techniques is reasonable. Of note that a lot of ICUs don't have bronchoscopy or ultrasound machines routinely available. Aim of this study was to describe a novel technique for safe blind percutaneous tracheotomy without assisting tools.

Patients and methods:

Enrolled patients were admitted to Critical Care Medicine Department in Alexandria University Hospitals in the period from 1st January 2018 to 31st December 2021. Approval of the Medical Ethics Committee of Alexandria Faculty of Medicine was obtained. An informed consent was taken from the patients' next of kin before their enrollment in the study. All percutaneous tracheotomies were performed electively to intubated patients at the bedside. Inclusion criteria were adult patients ≥ 18 years indicated for tracheotomy. Exclusion criteria were obese patients with Body Mass Index (BMI) ≥ 45 kg/m2, severe coagulopathy, and unsuitable anatomy (e.g., previous cervical surgery, cervical trauma, or tumors).

Data collection on enrollment was age, sex, body mass index (BMI), neck circumference, and indication for tracheostomy. Patients were sedated (midazolam 1-2 mg and fentanyl 100-200 mcg), paralyzed (atracurium 0.5 mg/Kg), and monitored by mainstream capnography, pulse oximetry and noninvasive blood pressure. Synchronized Intermittent Mandatory Ventilation (SIMV) mode was used, and the ventilator set to deliver 6-8mL/kg tidal volume, respiratory rate 16/minute, and fraction of inspired oxygen (FiO2) 100% starting 15 minutes before and until 5 minutes after the completion of the procedure. Proper pre-procedural suctioning from both endotracheal tube and mouth cavity was done.

Guidewire dilating forceps (Grigges') technique was the method which has been applied during our work. Proper positioning: patient's neck was extended as much as possible by placing a rolled towel between the shoulder blades, the patient's neck and the bed were maintained in neutral position. The operative site was sterilized before draping with 10% povidone iodine solution. Lidocaine 2% was used as local anesthetic prior to beginning the intervention.

Transverse (1 cm) skin incision was made midway between the cricoid cartilage and the suprasternal notch, i.e., opposite the 2nd - 3rd or 3rd - 4th tracheal rings. Blunt dissection of subcutaneous fat and pre-tracheal tissue with mosquito clamp in a vertical direction was done till the tracheal rings were palpable.

Novel technique for safe blind airway access:

After palpating the trachea through the incision, a 14- G cannula over needle was advanced caudally into trachea piercing and penetrating the rigid anterior wall of the endotracheal tube. Success of airway access was sudden loss of resistance while protecting the posterior tracheal wall by the posterior wall of the endotracheal tube with the non-dominant hand fixing the trachea during the process.

Endotracheal piercing of needle was confirmed by aspirating air bubbles into the saline filled syringe attached to the cannula over needle. Caudally directed needle position will be changed during gradual withdrawal of the endotracheal tube to release the cannula over needle off the anterior wall of the endotracheal tube. By this time, the proximal end of the cannula over needle penetrating the ETT will have been changed its direction cranially.

Successful full withdrawal of the cannula over needle from the anterior wall of the endotracheal tube was tested by smooth caudal redirection of the cannula over needle without any readvancement of the endotracheal tube. Caudal redirection of the cannula over needle is a mandatory step to ensure subsequent free passage of the guidewire into the trachea.

Upon successful release of the proximal end of cranially directed cannula over needle from the ETT, deflation of the ETT cuff and caudal redirection was mandatory for subsequent free passage of the guidewire into the trachea. To prevent injuring the bared posterior tracheal wall by the sharp needle' s tip during caudal redirection, one mm withdrawal of the needle out of the plastic cannula was done to make its proximal end non-traumatizing.

Proper caudal placement of the cannula over needle into the tracheal lumen was reconfirmed by aspirating air bubbles into the saline filled syringe attached to the cannula over needle once more. The needle was then removed leaving the cannula in place. The J-guidewire was inserted through the caudally directed cannula into the trachea. Cannula was subsequently removed.

The rest of the procedure was continued as usual: A 14- G dilator was passed over the guidewire to start stoma formation in the anterior tracheal wall. The Grigges' (guidewire dilating forceps) was advanced along the wire until resistance was felt at the anterior tracheal wall. The forceps was opened, and the pre-tracheal tissues were dilated. The forceps was removed, reapplied to the guidewire, and readvanced until the jaws were passed through the anterior tracheal wall. Opening the forceps to dilate the anterior tracheal wall was carried out. The forceps was removed, and the tracheostomy tube was loaded on the introducer dilator and passed into the trachea through the dilated stoma.

At this point the flexible introducer and the guidewire were removed, the cuff was inflated, and the ventilation was switched from the ETT to the tracheotomy tube. The endotracheal tube was completely removed after adequate ventilation through tracheotomy tube. Ventilation was confirmed by end expiratory volume on the ventilator and auscultation of the patient. The tracheotomy tube was secured in place with a neck band, and a chest radiograph was performed.

Procedure time was recorded with a digital stopwatch, (two times were recorded: 1-Novel Technique Time (NT Time): time from tracheal tube puncture till J-guidewire insertion into the trachea & 2- Total Technique Time (TT Time): time from skin incision till tracheotomy tube insertion). Peri-procedural complications were recorded. They included procedure failure (with mentioning action taken to accomplish tracheotomy), cardiac arrest, bleeding (mention grades of bleeding), transient desaturation below 92%, false passage, and posterior tracheal wall injury. Furthermore, post-procedure chest radiograph was done to exclude pneumothorax, pneumomediastinum, and subcutaneous emphysema.

For safety purposes, bronchoscopy during the procedure was performed in the first twenty patients, to confirm midline tracheal puncture, changes in cannula over needle directions, integrity of the posterior tracheal wall, proper positioning of the guidewire, dilators, as well as tracheotomy tube while passing into the trachea.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for tracheostomy

Exclusion Criteria:

* Age <18, patients with severe coagulopathy, and unsuitable anatomy (e.g., previous cervical surgery, cervical trauma, or tumors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2021-12-19 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Percutaneous tracheostomy procedure | 7 days
  Novel technique time: which is the time from tracheal tube puncture till J-guidewire insertion into the trachea

SECONDARY OUTCOMES:
Complications of the procedure | 7 days
  Percentage of procedure failure Incidence of desaturation below 92 % Incidence of cardiac arrest Incidence of false passage Incidence of posterior tracheal wall injury Incidence of pneumothorax, pneumomediastinum and surgical emphysema

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Sharing will be provided when required
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after statistical analysis for one year
URL: http://med.alexu.edu.eg/portal/moodle/

REFERENCES:
- [Result] Ciaglia P, Firsching R, Syniec C. Elective percutaneous dilatational tracheostomy. A new simple bedside procedure; preliminary report. Chest. 1985 Jun;87(6):715-9. doi: 10.1378/chest.87.6.715. PMID 3996056
- See also: Main link — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&cad=rja&uact=8&ved=2ahUKEwiirOmmuo_3AhUPhv0HHWkDBy8QFnoECAUQAQ&url=https%3A%2F%2Fpubmed.ncbi.nlm.nih.gov%2F3996056%2F&usg=AOvVaw3rBgEgIRckoSouVrGcKkwP